CLINICAL TRIAL: NCT03799055
Title: Ultrasonography(Distance From Skin to Epiglottis) vs Conventional Methods (Mallampati Score & Thyromental Distance) for Prediction of Difficult Airway in Adult Patients
Brief Title: Ultrasonography vs Conventional Methods for Prediction of Difficult Airway in Adult Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Baher Said Elshahat Mohamed Abdelhady, Principal investigator, Benha University
Other Study IDs: Us in difficult airway
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- easy intubation: Cormack _Lehane : 1&2
- difficult intubation: Cormack _Lehane : 3&4

SUMMARY:
The aim of this study to assess and compare between methods of prediction of difficult airway including Mallmpati score , thyromental distance and us measured distance from skin to epiglottis(DES) t the level of thyrohyoid membrane in adult patients requiring endotracheal intubation for an elective surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesia class 1,2and 3.
* elective surgical procedure requiring endotracheal intubation.
* Age 18_60 years old.
* BMI less than 40kg/meter square.

Exclusion Criteria:

* patients refusal.
* Unable to give consent.
* Preexisting airway malformations or pathology.
* History of difficult intubation.
* Pregnancy.
* Patients with tracheostomy tube.
* BMI more than 40 kg/meter square.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients at Benha University Surgical Hospital scheduled for elective surgical procedures requiring endotracheal tube
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Prediction of difficult airway | Preoperative
  Assess which method is better for prediction of difficult airway DES or conventional

CONTACTS AND LOCATIONS:
Overall Officials: Faculty Of Medicine, Study Director — faculty of medicine
Locations (1):
- Benha University Hospital, Banhā, Banha, Egypt

IPD SHARING:
Plan to Share IPD: No